CLINICAL TRIAL: NCT03506503
Title: Condensed Nanofat Grafting for Treatment of Androgenetic Alopecia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinan University Guangzhou (Other)
Responsible Party: Principal Investigator, Hongwei Liu, professor, Jinan University Guangzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019004
Record Dates: First submitted 2018-04-14; First posted 2018-04-24 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Androgenic Alopecia
Keywords: nanofat; hair loss; prp
MeSH Terms: conditions — Alopecia; Insomnia, Fatal Familial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- processed Nanofat grafting (Experimental): processed autologous Nanofat will be injected into the area of the scalp with androgenic alopecia.
  Interventions: Procedure: Nanofat grafting

INTERVENTIONS:
Procedure: Nanofat grafting — hair loss area will be treated by processed autologous Nanofat grafting

SUMMARY:
Nowadays, multiple treatment modalities have been applied clinically to treat androgenic alopecia, such as Follicular unit transplantation(FUT), finasteride, platelet-rich plasma injection(PRP), etc. In this clinical trial, the investigators aim to analyze the effect of nanofat grafting on treating androgenic alopecia in male.

DETAILED DESCRIPTION:
The investigators will treat the hair loss area of a patient by processed nanofat grafting. The participants were asked to come back 1、3、6、9、12 months after treatment for further follow-up.

Before and after the treatment, the hair and follicular will be assessed subjectively by satisfaction assessment, dermatoscope.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with androgenic alopecia aging from 18 to 50.
* No scars and wounds on the alopecia area.
* No skin disease or serious cardiovascular disease.
* Preoperative examinations remain healthy.

Exclusion Criteria:

* Serious chronic heart, liver, kidney, blood system disease
* Allergic diseases, skin inflammation or wounds
* Alopecia but not androgenic alopecia
* Acute or chronic infection
* Take anticoagulant drugs
* Active vitiligo, psoriasis, systemic lupus erythematosus

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Dermatoscope | Baseline and at1,3,6,9,12 months after the treatment
  the density of hair follicle and diameter of hair will be analized by dermatoscope before and after the treatment of Nanofat grafting.

OTHER OUTCOMES:
Satisfaction assessments | 1,3,6,12 months after treatment
  the satisfaction will be assessed after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonnard P, Verpaele A, Peeters G, Hamdi M, Cornelissen M, Declercq H. Nanofat grafting: basic research and clinical applications. Plast Reconstr Surg. 2013 Oct;132(4):1017-1026. doi: 10.1097/PRS.0b013e31829fe1b0. PMID 23783059
- [Background] Won CH, Park GH, Wu X, Tran TN, Park KY, Park BS, Kim DY, Kwon O, Kim KH. The Basic Mechanism of Hair Growth Stimulation by Adipose-derived Stem Cells and Their Secretory Factors. Curr Stem Cell Res Ther. 2017;12(7):535-543. doi: 10.2174/1574888X12666170829161058. PMID 28875863
- [Background] Gu Z, Li Y, Li H. Use of Condensed Nanofat Combined With Fat Grafts to Treat Atrophic Scars. JAMA Facial Plast Surg. 2018 Mar 1;20(2):128-135. doi: 10.1001/jamafacial.2017.1329. PMID 28975248